CLINICAL TRIAL: NCT02802930
Title: A Randomized Study to Assess the Potential for Phototoxicity of SPF 50 Y65 110, SPF 50 Y51 002 and SPF 15 V27-104 in Human Subjects
Brief Title: Test the Phototoxicity of Sunscreen Products
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: 18287
Record Dates: First submitted 2016-06-14; First posted 2016-06-16 (Estimated); Last update posted 2018-12-12 (Actual); Status verified 2018-12

CONDITIONS: Sunscreen Agents
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SPF 50 Y65 110, SPF 50 Y51 002, and SPF 15 V27 104 (Experimental): All test products (SPF 50 Y65 110,SPF 50 Y51 002, and SPF 15 V27 l 04 compared to that of a negative control [0.9% NaCl]) were tested simultaneously on each subject.
  Interventions: Drug: SPF 50 Y65 110 (BAY987519); Drug: SPF 50 Y51 002 (BAY987519); Drug: SPF 15 V27 104 (BAY987519); Drug: Sodium chloride [NaCl]

INTERVENTIONS:
Drug: SPF 50 Y65 110 (BAY987519) — Application of 200 µL in an occlusive patch of Webril (0.150 ± 0.010 mg) compared to that of a negative control (0.9% sodium chloride, NaCl) and followed by irradiation with UV A and UVB.
Drug: SPF 50 Y51 002 (BAY987519) — Application of 200 µL in an occlusive patch of Webril compared to that of a negative control (0.9% sodium chloride, NaCl) and followed by irradiation with UV A and UVB.
Drug: SPF 15 V27 104 (BAY987519) — Application of 200 µL in an occlusive patch of Webril compared to that of a negative control (0.9% sodium chloride, NaCl) and followed by irradiation with UV A and UVB.
Drug: Sodium chloride [NaCl] — Negative control (200 µL, 0.9% sodium chloride [NaCl]) after a single 24 h application of test materials followed by irradiation with ultraviolet A (UVA) and ultraviolet B (UVB).

SUMMARY:
The primary objective of this study was to evaluate the potential for phototoxicity of the sun care products SPF 50 Y65 110, SPF 50 Y51 002, and SPF 15 V27 104 compared to that of a negative control (0.9% sodium chloride [NaCl]) after a single 24 h application of test materials followed by irradiation with ultraviolet A (UVA) and ultraviolet B (UVB).

The secondary objective of this study was to evaluate the safety of the sun care products SPF 50 Y65 110, SPF 50 Y51 002, and SPF 15 V27 104 combined with UVA/B irradiation by monitoring adverse events (AEs) throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, aged 18 to 65 years
* Good general health, as assessed by medical history and brief visual examination of the skin
* Fitzpatrick skin Type I IV, determined by interview at screening
* Willing and able to practice an acceptable measure of contraception during the study, if female of childbearing potential
* Willing to follow study rules, which include: no sun exposure; avoidance of activities that would cause excessive sweating; and no use of lotions, creams, or oils on the back area
* Must be willing not to change current brand of personal care products such as soaps, body washes, laundry detergent, body sprays, and body spritzes while participating in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-04-20 (Actual); Primary Completion 2015-04-26 (Actual); Study Completion 2015-04-26 (Actual)

PRIMARY OUTCOMES:
Skin irritation | up to 1 week
  Skin irritation was rated on a scale from 0-7 where 0 is no evidence of irritation and 7 is strong reaction spreading beyond test site

SECONDARY OUTCOMES:
Number of adverse event as a measure of safety and tolerability | up to 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Pinellas Park, Florida, United States